CLINICAL TRIAL: NCT00263562
Title: Randomized Trial of High-dose Intravenous Methylprednisolone and Steroid Taper for Vaso-occlusive Crises in Sickle Cell Disease
Brief Title: Steroid Treatment for Sickle Cell Pain Crisis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor enrollment, availability of more effective medications
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Andrea Cruz, Associate Professor, Pediatrics-Emergency Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-17689
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
Keywords: Sickle cell disease; vaso-occlusive crisis; steroid treatment
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Steroid arm (Experimental): Receipt of methyprednisolone pulse dose: 15mg/kg to a maximum of 1 gram; following this, the patients also received a steroid taper with oral prednisone:Day 2: Prednisone 2mg/kg PO BID Day 3: Prednisone 2mg/kg PO daily Day 4: Prednisone 1mg/kg PO daily Day 5: Prednisone 1mg/kg PO daily
  Interventions: Drug: Steroid arm
- Comparison Group (Placebo Comparator): Patients receiving usual care, with receipt of placebo (saline in lieu of intravenous methylprednisolone infusion or a number of placebo pills equivalent in number to what would have been received for the prednisone.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Steroid arm — Day 1: Solumedrol 15 mg/kg (maximum 1 gram) Day 2: Prednisone 2mg/kg PO BID Day 3: Prednisone 2mg/kg PO daily Day 4: Prednisone 1mg/kg PO daily Day 5: Prednisone 1mg/kg PO daily
  Other Names: Systemic corticosteroid receipt
  Arms: Steroid arm
Other: Placebo — Patients received normal saline in lieu of intravenously-administered methylprednisolone and placebo pills equal in number to the steroid pills received in the steroid arm
  Arms: Comparison Group

SUMMARY:
The painful episode is the most common problem experienced by children with sickle cell disease. Although various treatments are available during painful episodes, the medication most commonly given for pain is a pain medication such as morphine. Fluids are also used. Even with these treatments, many children still have severe pain that is difficult to control. In addition to pain medications, there are other medications that may be useful. Methylprednisolone (solumedrol) and prednisone are a group of medications called steroids that may be helpful for painful episodes. These medications are known to lower the amount of inflammation (this means swelling, tenderness, and soreness) in the body. Because this medication may help with your pain, you are being asked to be a part of this study. These types of medications are used in other illnesses such as asthma, especially during times when the illness has gotten worse.

The main purpose of this study is to see if the methylprednisolone and prednisone will lower the amount of pain and the length of hospital stay.

In addition to the pain medication you will normally receive, you will be assigned to one of 2 groups: 1) the experimental group with the active form of the medicine, or 2) a comparison group without the active form of the medicine. In either group, you will still receive all of the treatments you would normally receive for a painful episode, including pain medicines and fluids. You and your doctors will not know what group you will be assigned.

If you decide to be a part of the study the following will happen:

For the first 5 days, you will be asked to: 1) describe your current pain (0=no pain to 10=a lot of pain), worst pain (0=no pain to 10=a lot of pain), least pain (0=no pain to 10=a lot of pain), and the amount of pain relief (0=no relief to 10=complete relief); 2) describe any signs or symptoms you feel, including filling out a pain scale form each day; 3) and take the medicines for 5 days, either at home or when in the hospital. Thirty days after the study, a study researcher will call and will ask questions about your pain, any painful episodes, and any medications you had. If you are discharged home sooner than 5 days after the start of the study, research staff will call you to ask you these questions, remind you to fill out your pain forms, and remind you to take your medicine. If you are discharged home, you will be given pain scales to fill out each day at home.

DETAILED DESCRIPTION:
In the United States, 9% of African Americans have sickle cell trait and 1 in 600 has sickle cell disease. Vaso- occlusive crises in sickle cell disease remain a frequent cause of severe pain, leading to emergency room visits, hospitalizations, and dependence upon narcotics for analgesia. Current treatments for vaso-occlusive crises includes IV analgesia with narcotics, NSAIDS, and hydration. Admissions can be frequent, prolonged, and can significantly diminish quality of life.

Understanding the pathophysiology of vaso-occlusive crises helps to find possible treatments. The etiology of vaso- occlusive crises includes HbS polymerization; sickle erythrocyte polymerization; endothelial damage; and inflammation, reperfusion injury, and oxidant radical production (Steinberg et al, Hematology, 2004). For example, hydroxyurea works by increasing the amount of fetal hemoglobin (HbF) and thus inhibiting polymerization, and reduces the incidence of pain by nearly 50%. Glucocorticoids would be expected to exert effects on the endothelium and inflammation.

Vaso-occlusive crises share similar features with other inflammatory processes, including clinical symptoms of swelling, erythema, and warmth; and laboratory findings of leukocytosis and elevated ESR. It has previously been theorized that glucocorticoids, which are used in many other inflammatory disorders, could decrease the duration or severity of vaso-occlusive crises. Methylprednisolone is a corticosteroid which decreases inflammation by suppression of migration of polymorphonuclear leukocytes and reversal of increased capillary permeability (Takemoto, et al 2004). A randomized, placebo-controlled study of 2 doses of intravenous methylprednisolone for vaso-occlusive crisis showed that the duration of severe pain and the need for inpatient analgesia was decreased in patients who received methylprednisolone; however the intervention patients had more rebound attacks than those who received placebo. (Griffin et al, NEJM, 1994)

Previous studies have examined long-term administration of steroid hormones including testosterone, progesterone, and medroxyprogesterone to patients with sickle cell disease. In placebo-controlled crossover trials, patients who received steroids had fewer vaso-occlusive episodes than placebo-treated patients (Isaacs et al, Lancet,1972; DeCeulaer et al, Lancet, 1982). Initial reports of glucocorticoids for vaso-occlusive crisis include an uncontrolled report of hydrocortisone as adjunctive therapy for VOC (Araujo et al, Blood, 1990). A case report showed efficacy of dexamethasone for vaso-occlusive crisis in children (Robinson et al, Lancet, 1979). The mechanism of steroids effect is uncertain.

In acute chest syndrome, which shares many clinical features with vaso-occlusive crises, intravenous therapy with dexamethasone has been shown to reduce the length of hospital stay, prevent clinical deterioration, and reduce the need for blood transfusion (Bernini et al, Blood, 1998).

In a placebo-controlled trial of high-does methylprednisolone for VOC, patients with severe pain requiring hospital admission were randomized to receive methylprednisolone or placebo (15 mg/kg to maximum 1 gram) at admission and again 24 hours later. The duration of inpatient analgesia was significantly shorter in patients who received methylprednisolone. However, patients who received methylprednisolone were much more likely to be readmitted shortly after finishing therapy. In addition, the study was criticized because patients did not rate their pain, and very few patients received patient-controlled analgesia while hospitalized.

Since this trial was published, there have been other advances in the standard management of VOC. Ketorolac, a non-steroidal analgesic, is now a standard adjunctive therapy, and most patients are quickly placed on patient-controlled analgesia. In addition, more patients now receive chronic, preventative therapies such as hydroxyurea and chronic transfusions.

We are therefore interested in repeating and expanding upon the results obtained several years ago and in evaluating the role of steroids if given over a slightly longer period of time.

The primary objective of this study is to determine whether the use of high-dose methylprednisolone followed by steroid taper decreases the duration of hospitalization and severity of pain in VOC of sickle cell disease.

Primary Hypothesis: The experimental group treated with high-dose methylprednisolone and steroid taper plus conventional therapy will have an improvement in pain scores using a 10-point scale.

In addition, the secondary objectives were:

1. duration of inpatient admissions
2. to examine the number and type of complications and side effects (infection, hypertension, and GI bleeding)
3. to determine rate of recurrent episodes of pain within one month of treatment.
4. to determine whether the amount of analgesic used will decrease during the hospitalization, as measured by the # of days in which IV opioids were given.

ELIGIBILITY:
Inclusion Criteria:

Sickle cell and acute pain Age 8 and up English or Spanish-speaking

Exclusion Criteria:

Fever greater than 101 Acute chest syndrome or pneumonia Other SS complications (sequestration, aplastic crisis) Other explanation for pain (chronic, AVN, surgical) History of GI bleeding, HTN, or hyperglycemia/DM

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2008-06-13 (Actual); Study Completion 2008-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention (Steroids): Day 1: Solumedrol 15 mg/kg (maximum 1 gram) Day 2: Prednisone 2mg/kg PO BID Day 3: Prednisone 2mg/kg PO daily Day 4: Prednisone 1mg/kg PO daily Day 5: Prednisone 1mg/kg PO daily
- Placebo: a comparison group who received standard of care therapy for acute chest syndrome, with normal saline substituted in lieu of IV solumedrol (methylprednisolone) and placebo pills in lieu of prednisone tablets (same # of tablets of placebo given as would have been administered to the intervention arm).
Period: Overall Study
Arm/Group | Intervention (Steroids) | Placebo
Started (This study was terminated early and not completed.) | 9 | 9
Completed | 6 | 9
Not Completed | 3 | 0
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm: Receipt of IV pulse of steroids (methylprednisolone) followed by a steroid taper on the subsequent days: Day 2: Prednisone 2mg/kg PO BID Day 3: Prednisone 2mg/kg PO daily Day 4: Prednisone 1mg/kg PO daily Day 5: Prednisone 1mg/kg PO daily
- Placebo Arm: Receipt of usual care, with administration of placebo: 1) normal saline in lieu of IV methylprednisolone followed by 2) placebo tablets in lieu of prednisone tablets.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Placebo Arm | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 6.5 [4.9 to 8.2] | 10.6 [7.3 to 13.2] | 9.6 [6 to 12.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Severity of pain using a 10-point scale ranging from 1-10, with higher numbers corresponding to worsening pain.
Time Frame: 30 days
Population: Analyzed by intent to treat (ITT), with the 3 protocol deviations in the intervention arm (all 3 received placebo) counting toward the intervention arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Intervention (Steroids): Receipt of pulse IV dose of methylprednisolone followed by a tapering dose of systemic oral corticosteroids (prednisone).
- Placebo Group: Receipt of usual care, with normal saline in lieu of IV methylprednisolone and placebo tablets in lieu of prednisone tablets.
Arm/Group | Intervention (Steroids) | Placebo Group
Number analyzed (Participants) | 9 | 9
score on a scale | 4.3 [2.5 to 6.7] | 4.5 [2.1 to 7.1]

2. Secondary Outcome: Duration of Hospitalization
Description: Length of stay (from emergency department arrival to discharge from the inpatient unit), in days, through hospitalization, up to 15 days
Time Frame: Through hospitalization, up to 15 days
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Steroid Arm | Comparison Group
Number analyzed (Participants) | 9 | 9
days | 6.5 [4.9 to 8.2] | 10.6 [7.3 to 13.2]

3. Secondary Outcome: Number of Participants With Complications and Adverse Events
Description: To describe adverse events, including infection, hypertension, and/or GI bleeding
Time Frame: 30 days
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Arm | Comparison Group
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Recurrent Episodes of Pain Within 1 Month of Treatment
Description: Number of recurrent episodes of pain within 1 month of treatment
Time Frame: 30 days
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Arm | Comparison Group
Number analyzed (Participants) | 9 | 9
Participants | 0 | 1

5. Secondary Outcome: Number of Days Analgesia Used
Description: # of days during which the child received parenterally-administered opioids through hospitalization, up to 15 days.
Time Frame: Through hospitalization, up to 15 days
Population: Intent to treat
Measure: Median (Full Range); unit: days
Arm/Group | Steroid Arm | Comparison Group
Number analyzed (Participants) | 9 | 9
days | 4 [1 to 7] | 3 [1 to 8]

ADVERSE EVENTS:
Groups:
- Intervention Arm (Steroids): Receipt of IV followed by oral systemic corticosteroids
- Control Group: Standard care for acute chest syndrome, with normal saline used in lieu of IV methylprednisolone and placebo tablets used in lieu of oral steroid tablets.
Arm/Group | Intervention Arm (Steroids) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No